CLINICAL TRIAL: NCT06647329
Title: CAR-T Technology for the Treatment of Recurrent/Refractory Malignant Hematological and Lymphatic Tumors: Multi-Center Clinical Study on Safety and Efficacy
Brief Title: CAR-T Technology for Recurrent/Refractory Malignant Hematological and Lymphatic Tumors
Acronym: CAR-T Therapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital Investigator Affiliation, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblCAR-T
Record Dates: First submitted 2024-10-10; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: CAR-T Cell Therapy; Lymphomas
Keywords: CAR-T therapy; Recurrent/Refractory Malignant Hematological Lymphomas
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): CAR-T therapy
  Interventions: Biological: CAR-T Therapy

INTERVENTIONS:
Biological: CAR-T Therapy — CAR-T Technology for the Treatment of Recurrent/Refractory Malignant Hematological Lymphomas

SUMMARY:
evaluate the safety and Esfficacy of CAR-T technology for the treatment of recurrent/refractory malignant hematological lymphomas

DETAILED DESCRIPTION:
Patients with recurrent/refractory malignant hematological lymphomas were treated with CAR-T technology

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet all of the following conditions to be included:

1. The participant has given informed consent and signed the consent form, and is willing and capable of complying with the scheduled visits, study treatment, laboratory examinations, and other trial procedures.
2. Clinically diagnosed as having relapsed/refractory malignant hematologic tumors:

   2.1 Diagnosed as CD19+ and/or CD20+ and/or CD22+ B-cell tumors through pathological and histological examinations, and the participant meets the criteria for relapsed or refractory B-cell malignancies as follows:

   B-cell tumors include the following three categories:

   A. B-cell acute lymphoblastic leukemia (B-ALL); B. Indolent B-cell lymphomas (CLL, FL, MZL, LPL, HCL); C. Aggressive B-cell lymphomas (DLBCL, BL, MCL).

   2.1.1. Refractory/relapsed B-cell leukemia (meeting one of the following four criteria): A. Relapse within 6 months after initial remission; B. Initial refractory after 2 cycles of standard chemotherapy without achieving complete remission; C. Relapse or refractory after first-line or multi-line salvage chemotherapy without achieving complete remission; D. Not suitable for hematopoietic stem cell transplantation, or have abandoned transplantation due to conditions, or relapse after transplantation.

   2.1.2. Refractory/relapsed B-cell lymphoma (meeting one of the first four criteria plus the fifth): A. Tumor shrinkage of less than 50% or disease progression after 4 cycles of standard chemotherapy; B. Achieved CR after standard chemotherapy, but relapsed within 6 months; C. Relapsed 2 times or more after achieving CR; D. Not suitable for hematopoietic stem cell transplantation, or have abandoned transplantation due to conditions, or relapse after transplantation;

   E. The participant must have received sufficient prior treatment, including at least:
   1. Anti-CD20 monoclonal antibodies
   2. Combination chemotherapy containing anthracyclines.

   2.2 Refractory/relapsed multiple myeloma: Progressed after at least 3 lines of treatment (at least one proteasome inhibitor and one immunomodulator used).

   2.3 Presence of measurable or evaluable lesions: A. For lymphoma patients, a single lesion ≥15 mm or two or more lesions ≥10 mm, or PET-positive lesions determined according to Lugano criteria; B. For leukemia and myeloma patients, bone marrow MRD must be persistently positive or positive relapse.
3. Age 14-75 years (inclusive), both male and female.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Treatment-related antigen test results must be positive:

   A. For lymphoma: CD19/CD20/CD22 (immunohistochemical results positive within six months); B. For acute lymphoblastic leukemia: CD19/CD22 (tumor cells detected positive by flow cytometry in bone marrow at screening, or extramedullary lesions with positive immunohistochemistry results within six months); C.For multiple myeloma: BCMA (tumor cells detected positive by flow cytometry in bone marrow at screening, or extramedullary lesions with positive immunohistochemistry results within six months).
6. Expected survival time greater than 3 months from the date of signing the informed consent form.
7. HGB ≥ 70 g/L (transfusion allowed).
8. Liver and kidney function, and cardiopulmonary function must meet the following requirements: a) Creatinine ≤ 1.5 × ULN; b) Left ventricular ejection fraction ≥ 50%; c) Blood oxygen saturation > 90%; d) Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN.
9. Participants with a plan for pregnancy must agree to use contraception before enrollment and for six months after the study begins; if the participant becomes pregnant or suspects pregnancy, they must immediately notify the investigator.

Exclusion Criteria:

Participants who meet any of the following conditions are not eligible for inclusion:

1. History of any of the following cardiovascular diseases within the past 6 months: New York Heart Association (NYHA) class III or IV heart failure, cardiovascular intervention (angioplasty or stenting), myocardial infarction, unstable angina, or other clinically significant heart diseases.
2. History of severe pulmonary dysfunction.
3. Concurrent advanced malignant tumors.
4. Concurrent systemic fungal, bacterial, viral, or other infections that cannot be effectively controlled.
5. Concurrent severe autoimmune diseases or congenital immunodeficiency.
6. Active hepatitis (positive HBV DNA or HCV RNA testing).
7. Human Immunodeficiency Virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection.
8. History of severe allergic reactions to biologics (including antibiotics).
9. Less than 6 months since undergoing allogeneic hematopoietic stem cell transplantation.
10. Acute or chronic graft-versus-host disease (GvHD).
11. History of deep vein thrombosis (DVT) (cancer-related thrombosis) or pulmonary embolism (PE) within 3 months prior to signing the informed consent form.
12. Anticoagulation treatment for DVT or PE within 3 months prior to signing the informed consent form.
13. History or clinical significance of CNS diseases at screening, such as epilepsy, seizure disorders, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or mental disorders.
14. Pregnant or breastfeeding women. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to the start of lymphocyte-depleting chemotherapy.
15. Use of any of the following medications or treatments within the specified time before leukapheresis:

    A. Use of alemtuzumab within the past 6 months prior to leukapheresis; B. Use of anti-CD20 monoclonal antibodies within 7 days prior to leukapheresis; C. Use of Venetoclax within 4 days prior to leukapheresis; D. Use of lenalidomide within 3 days prior to leukapheresis; E. Use of Idelalisib within 2 days prior to leukapheresis; F. Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent > 20 mg/day) within 7 days prior to leukapheresis or 72 hours prior to CAR-T administration. However, physiological replacement, topical, and inhaled steroids are permitted; G. Use of investigational drugs within 4 weeks prior to leukapheresis. However, if treatment was ineffective or the disease progressed during the trial and at least 3 half-lives have elapsed before leukapheresis, enrollment is allowed; H. Received donor lymphocyte infusion (DLI) within 6 weeks prior to CAR-T administration.
16. Any factors judged by the investigator that may affect compliance with the study protocol, including uncontrollable medical, psychological, familial, sociological, or geographical factors, or unwillingness or inability to comply with the required procedures of the study protocol.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | 6 months
  evaluate the efficacy of CAR-T cell infusion for the treatment of relapsed/refractory malignant hematological tumors

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided